CLINICAL TRIAL: NCT02984722
Title: Extended-release vs Immediate-release Metformin in PCOS Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Metformin XR
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

ARMS (2):
- 1 (Experimental): PCOS women treated with 1500 mg/die of extended-release metformin
  Interventions: Drug: Metformin
- 2 (Experimental): PCOS women treated with 1500 mg/die of immediate-release metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
The aim of our study is to compare the different effects of 6 months treatment with extended-release metformin and immediate-release metformin on clinical, endocrine and metabolic parameters in women affected by polycystic ovary syndrome. We also evaluate gastrointestinal disorders associated with the two different compouds.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS in accordance with Rotterdam criteria

Exclusion Criteria:

* pregnancy
* diabetes mellitus (or impaired glucose tolerance as determined by a standard 75 gr oral glucose tolerance test)
* past history of cardiovascular diseases
* past history of gastro-intestinal diseases
* significant liver or renal dysfunction (hypothalamic, pituitary, thiroidal or adrenal);
* neoplasms.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Gastro intestinal disorders | 6 months

SECONDARY OUTCOMES:
number of cycles in 6 months of therapy | 6 months
insulin levels | 6 months
hirsutism score | 6 months
androstenedione levels | 6 months
testosterone levels | 6 months
free androgen index | 6 months
dheas levels | 6 months
ovarian volume | 6 months
total cholesterol | 6 months
tryglycerides levels | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of Sacred Heart, Rome, Rome, Italy